CLINICAL TRIAL: NCT07396389
Title: Modèle de Performance Subjective Généralisé
Brief Title: Understanding How Young Adults Perceive Blurred Image Quality and Creating a Model Predicting Their Quality Ratings
Acronym: GESUVIPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WS10490; 2025-A02625-44 (Other: ANSM RCB)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Young Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): young adults that are provided with simulated images to be observed and rated
  Interventions: Device: eye exam; Other: image rating

INTERVENTIONS:
Device: eye exam — participants will follow a complete eye exam
Other: image rating — participants will have to rate the perceived quality of images on a 10 points scale

SUMMARY:
This clinical study wants to understand how blurred images look to young adults.

The main question is: How do different kinds of images and different kinds of blur change the way people think those images look? Participants will get an eye exam, then look at several blurred images and rate how good or bad each one looks on a quality scale from 1 (very bad) to 10 (very good).

ELIGIBILITY:
Inclusion Criteria:

* Distance refractive error (equivalent sphere) between -7 D and +5 D
* Astigmatism below 4D
* Minimum corrected visual acuity: 10/10

Exclusion Criteria:

* Aphakic or pseudophakic eye surgery
* Reported systemic pathology that affects vision
* Medical treatment or taking medications that affect vision
* Severe ocular pathology declared, involving a loss of visual field as in glaucoma, a loss of acuity
* Reported neurological deficit, including a history of seizure or sensorimotor coordination disorders, vestibular or cerebellar pathology
* Binocular vision problems such as amblyopia, strabismus, or double vision

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Subjective image quality rating on a quality scale from 1 (very bad) to 10 (very good) | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- LABORATOIRE LuMIn - ENS Paris-Saclay, Gif-sur-Yvette, France

IPD SHARING:
Plan to Share IPD: No